CLINICAL TRIAL: NCT03455855
Title: Prospective, Non-randomized, Multicenter Clinical Study of the JETSTREAM™ Atherectomy System (Jetstream) in Treatment of Occlusive Atherosclerotic Lesions in the Superficial Femoral and/or Proximal Popliteal Arteries in Chinese Patients
Brief Title: Jetstream in Treatment of Occlusive Atherosclerotic Lesions in the SFA and/or PPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6050
Record Dates: First submitted 2018-02-24; First posted 2018-03-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerosis
Keywords: Atherectomy; occlusive atherosclerotic lesions
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- treated with the Jetstream System (Experimental): It is intended that all patients with qualifying lesions would be considered for enrollment and treated with the Jetstream System.
  Interventions: Device: Jetstream System

INTERVENTIONS:
Device: Jetstream System — including Atherectomy Console (Jetstream Console) and Atherectomy Catheter(Jetstream Catheter), intended for use in atherectomy of the peripheral vasculature and to break apart and remove atherosclerotic disease, debris, and thrombus from the SFA and/or PPA.

SUMMARY:
This clinical study is a prospective, non-randomized, multicenter, single-arm study to demonstrate the acceptable safety and performance of the JETSTREAM™ Atherectomy System (Jetstream) used during percutaneous peripheral vascular intervention in patients with occlusive atherosclerotic lesions in the native SFA and/or PPA. It is intended that all patients with qualifying lesions would be considered for enrollment and treated with the Jetstream System.

DETAILED DESCRIPTION:
study objectives: To evaluate the safety and effectiveness of JETSTREAM™ Atherectomy System (Jetstream) for treating symptomatic Chinese patients with occlusive atherosclerotic lesions in native superficial femoral artery (SFA) and/ or proximal popliteal arteries (PPA)during percutaneous peripheral vascular intervention.

Planed Indications for use: The Jetstream System is intended for use in atherectomy of the peripheral vasculature and to break apart and remove atherosclerotic disease, debris, and thrombus from the SFA and/or PPA.

Primary Safety Endpoint: Major Adverse Event (MAE), defined as all-cause death, target limb unplanned major amputation and/or target lesion revascularization (TLR), within 30 days post index procedure

Primary Effectiveness Endpoint: Acute reduction of percent diameter stenosis (%DS) post atherectomy but prior to any adjunctive therapy, when compared to its baseline diameter stenosis (absolute mean percentage).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older
2. Subject or the subject's legal representative is willing and able to provide consent before any study-specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits
3. Subject has documented chronic, symptomatic lower limb ischemia defined as Rutherford categories 2 - 4, and is eligible for percutaneous peripheral vascular intervention
4. Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA, and meet all of following angiographic criteria by visual assessment:

   i. Atherosclerotic lesion with diameter stenosis ≥70% ii. Guidewire must cross lesion(s) within the true lumen, without a sub-intimal course by physicians performed, based on visual estimate iii. Minimum vessel diameter proximal to the lesion ≥ 3 mm and < and =6 mm iv. Lesion length of single or multiple focal stenosis or chronic total occlusion (CTO) lesion can be up to 15 cm long v. Target lesion located at least 3 cm above the inferior edge of the femur
5. Patent infrapopliteal and popliteal artery, i.e., single distal runoff or better with at least one of three vessels patent (< 50% stenosis by visual assessment) to the ankle or foot with no planned intervention

Exclusion Criteria:

1. Target lesion is located in the iliac artery or above the SFA
2. Target lesion stenosis < 70%
3. Target lesion is moderately to severely angulated (> 30°) or torturous at treatment segment
4. Target lesion/vessel previously treated with drug-coated balloon within 12 months prior to the index procedure
5. Target lesion/vessel previously treated with atherectomy, laser or other debulking devices prior to the index procedure
6. Target lesion/vessel with in-stent restenosis
7. Subjects who have undergone prior surgery or endovascular intervention of SFA/PPA in the target limb to treat atherosclerotic disease within 3 month prior to the index procedure
8. Use of drug-coated devices, or laser or any other debulking devices other than Jetstream System (such as CTO devices or cutting balloon) in the target limb during the index procedure
9. History of major amputation in the target limb
10. Documented life expectancy less than 12 months due to other medical co-morbid condition(s)
11. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated
12. Known history of coagulopathy or hypercoagulable bleeding disorder
13. Known hypersensitivity/allergy to the investigational devices or protocol related therapies (e.g., nitinol, stainless steel or other stent materials, and antiplatelet, anticoagulant, thrombolytic medications)
14. Platelet count < 80,000 mm3 or > 600,000 mm3 or history of bleeding diathesis
15. Undergoing hemodialysis or concomitant renal failure with a serum creatinine > 2.0 mg/dL (176.8umol/L)
16. History of myocardial infarction (MI), stroke/cerebrovascular accident (CVA) or gastrointestinal bleeding within 6 months prior to the enrollment
17. Unstable angina pectoris at the time of enrollment.
18. History of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within past 14 days
19. Pregnant, breast feeding, or plan to become pregnant in the next 12 months
20. Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of enrollment or that clinically interferes with the current study endpoints (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies)
21. Septicemia at the time of enrollment
22. Presence of outflow lesions in the target limb requiring intervention during the index procedure
23. Presence of other hemodynamically significant lesions in the target limb requiring intervention within 30 days of enrollment
24. Acute ischemia and/or acute thrombosis of the target lesion/vessel prior to the index procedure
25. Presence of aneurysm in the target vessel
26. Perforated vessel as evidenced by extravasation of contrast media prior to the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2024-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 6 sites between Feb 2018 and Jan 2024. The first participant was enrolled on 5 Mar 2018 and the last participant was enrolled on 10 Jan 2023.
Pre-assignment Details: Approximately 80 subjects (including 20 roll-in subjects) in 10 sites planned to be enrolled. The sample of primary cohort is 60. The sample of roll in cohort depends on the site number. 2 roll-in subjects per site is required. Actually 6 site participated in this study, totally there are 72 subjects in all.
Groups:
- Primary Cohort: The overall sample size is consist of the primary cohort and roll-in subjects. A sample size of 60 subjects to be enrolled in the primary cohort at baseline.
- Roll in Cohort: The overall sample size is consist of the primary cohort and roll-in subjects. With additional 2 roll-in subjects per site and 6 sites are eligible for enrollment.
Period: Overall Study
Arm/Group | Primary Cohort | Roll in Cohort
Started | 60 | 12
Primary Endpoint(30days) | 60 | 12
Completed | 56 | 10
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Cohort | Roll in Cohort | Total
Number analyzed (Participants) | 60 | 12 | 72
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [45 to 86] | 64.9 [60 to 74] | 67.1 [45 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 50 | 7 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 12 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Effectiveness Endpoint-Acute Reduction of Percent Diameter Stenosis
Description: Acute reduction of percent diameter stenosis (%DS) post atherectomy but prior to any adjunctive therapy, when compared to its baseline diameter stenosis (absolute mean percentage).
Time Frame: Index Procedure (Core-lab will analysis the procedural angiograms to assess the acute reduction of percent diameter stenosis (%DS))
Population: 57/60 subjects from primary cohort and 11/12 subjects from roll in cohort received primary effectiveness endpoint analysis from core lab.
Measure: Mean (Standard Deviation); unit: percentage of DS(diameter stenosis)
Groups:
- Overall Cohort: The overall sample size is consist of the primary cohort and roll-in subjects.
Arm/Group | Primary Cohort | Roll in Cohort | Overall Cohort
Number analyzed (Participants) | 57 | 11 | 68
percentage of DS(diameter stenosis) | 39.3 (16.1) | 42.8 (11.1) | 39.9 (15.4)

2. Primary Outcome: The Primary Safety Endpoint-The Rate of Major Adverse Event (MAE) at 30 Days Follow up
Description: defined as all-cause death, target limb unplanned major amputation and/or target lesion revascularization (TLR), within 30 days post index procedure.
Time Frame: 30days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Cohort | Roll in Cohort | Overall Cohort
Number analyzed (Participants) | 60 | 12 | 72
Participants | 60 | 11 | 71

ADVERSE EVENTS:
Time Frame: 1 year
Description: MedDRA
Arm/Group | Primary Cohort | Roll in Cohort
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/12
Serious Adverse Events (participants affected / at risk) | 21/60 | 8/12
Other Adverse Events (participants affected / at risk) | 45/60 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort (N=60) | Roll in Cohort (N=12)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (12) | 3 (3)
Peripheral embolism (Vascular disorders) | 3 (3) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular wall hypertrophy (Vascular disorders) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Contrast media deposition (General disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort (N=60) | Roll in Cohort (N=12)
Peripheral artery stenosis (Vascular disorders) | 21 (21) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Vessel perforation (Vascular disorders) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 13 (13) | 8 (9)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Vascular stent restenosis (General disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03455855/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03455855/SAP_001.pdf